CLINICAL TRIAL: NCT05610683
Title: Comparison of the Removal of Uremic Toxins With Medium Cut-off and Super High-flux Vitamin E-coated Dialyzers The E-FLUX Randomized Study
Brief Title: Comparison of the Removal of Uremic Toxins With Medium Cut-off and Super High-flux Vitamin E-coated Dialyzers
Acronym: E-FLUX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Collaborators: Hemotech (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: E-FLUX
Record Dates: First submitted 2022-10-27; First posted 2022-11-09 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-04

CONDITIONS: End Stage Renal Disease (ESRD)
Keywords: super high-flux hemodialysis; medium cut-off hemodialysis; beta2-microglobulin
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Intervention Model Description: The E-FLUX is a prospective randomized open-label cross over study. The study will include 38 patients established on HF-HD randomly assigned to receive either 3 months of SHFVE-HD followed by 3 months of MCO-HD, or vice versa.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SHFVE-HD group (Experimental): Hemodialysis sessions using the VieX™ (Polysulfone, surface area: 2.1 m², sterilization gamma, ultrafiltration coefficient: 104.3 ml/h/mmHg, Asahi Kasei Medical, Japan).
  Interventions: Device: Hemodialysis sessions using SHFVE dialyzer (VieX™) or the MCO (Theranova 500™) dialyzer
- MCO-HD group (Experimental): Hemodialysis sessions using the Theranova 500™ (Baxter healthcare Corporation Deerfield, USA; surface area 2 m², ultrafiltration coefficient: 59 ml/h/mmHg).
  Interventions: Device: Hemodialysis sessions using SHFVE dialyzer (VieX™) or the MCO (Theranova 500™) dialyzer

INTERVENTIONS:
Device: Hemodialysis sessions using SHFVE dialyzer (VieX™) or the MCO (Theranova 500™) dialyzer — Patients will receive thrice weekly 4 hours hemodialysis sessions during 3 months

SUMMARY:
End-stage renal disease (ESRD) induces an accumulation of uremic toxins responsible for increased morbidity and mortality. These toxins cover a wide range of molecules, classified according to their molecular weight as small-size (< 500 Da), middle-size (500 Da-60 kDa), and protein-bound toxins.

Specific complications have been associated with the accumulation of middle-size toxins, including beta2-microglobulin (12 kDa), myoglobin (17 kDa), prolactin (23 kDa), alpha1-microglobulin (33 kDa), alpha1-glycoprotein (44 kDa), kappa (22 kDa) and lambda (45 kDa) free light chains (FLC). Moreover, mediators of oxidative stress such as asymmetric dimethylarginine, malondialdehyde, oxidative-LDL and inflammatory cytokines such as Interleukin-6 (IL)-6, IL1-β, TNF-α have been involved in atherosclerosis, malnutrition, cardiovascular events and mortality.

Hemodialysis (HD) remains the main standard modality of renal replacement therapy in ESRD. In the past decade, low-flux hemodialysis was most commonly used, providing effective clearance of small solutes through diffusion, but negligible clearance of middle molecules. This limitation was insufficiently improved by the development of high-flux (HF) dialyzers due to their cut-off pores size values of approximately 15-20 kDa. In fact, most of middle molecules cannot be efficiently removed by HF-HD because of their molecular radii larger than that of membrane pores. Thus, HF dialyzers were used in post dilution on-line hemodiafiltration (OL-HDF) mode with high convection volumes and achieved greatest clearance of middle molecules. However, OL-HDF is generally not available in most HD centers and needs additional hardware technology. Therefore, several super high-flux (SHF) dialyzers integrating higher cut-off size pore value and achieving Beta2-microglobulin clearance > 70 ml/min were developed for HD mode. These SHF dialyzers used in HD (SHF-HD) provides similar middle molecules depuration compared to OL-HDF.

The recently developed medium cut-off (MCO) dialyzer (Theranova 500™, Baxter healthcare Corporation Deerfield, USA; surface area 2 m², ultrafiltration coefficient: 59 ml/h/mmHg) differs from conventional HF membranes by higher and controlled porosity resulting in a steep sieving curve with a cut-off value approaching that of albumin. MCO-HD has demonstrated efficient depuration of middle uremic toxins as compared to HF-HD, similar to that of OL-HDF. MCO-HD and SHF-HD are two new large pore size dialyzers currently used nowadays in HD.

In addition, the interaction between blood and membrane surface play a key role in generating oxidative stress and inflammation. Antioxidants such as vitamin E work by inhibiting LDL oxidation and by limiting cellular response to oxidized LDL. In HD patients, vitamin E may be integrated as a part of the HD procedure in the form of bioreactive dialysis membranes, in which the blood surface has been modified with alpha-tocopherol. Dialysis with vitamin E-coated membranes has been associated with an improvement in biocompatibility including circulating lipid peroxidation biomarkers and cytokine induction. In small studies, vitamin E coated dialyzers have been associated with reduced red blood count fragility and improvements in erythropoietin resistance index and erythropoietin requirements in HD.

VieX (Polysulfone, surface area: 2.1 m², sterilization gamma, ultrafiltration coefficient: 104.3 ml/h/mmHg, Asahi Kasei Medical, Japan), a novel SHF vitamin E-coated (SHVE) dialyzer, which has larger pore size than HF dialyzer, might provide higher middle molecules removal and biocompatibility improvement.

The aim of the present study was to compare the efficiency of the SHFVE dialyzer (VieX™) versus the MCO dialyzer (Theranova 500™) on the removal of beta2-microglobulin and other middle molecules in a non-inferiority fashion, and their respective effects on inflammation, oxidative stress and biocompatibility parameters.

DETAILED DESCRIPTION:
In a previous randomized study, it was found that compared to HF-HD after 3 months, MCO-HD was associated with higher middle molecules removal and significant decrease in beta2-microglobulin, oxidized low-density lipoprotein, kappa and lambda free light chain pre-dialysis levels, without change in other inflammatory and oxidative stress biomarkers. In addition, a modulation of inflammation has been demonstrated with MCO-HD in another randomized trial. After 3 months, MCO-HD was shown to downregulate the expression of the pro-inflammatory IL-6 and tumor necrosis factor (TNF) mRNA in peripheral leucocytes. Moreover, higher removal and decrease in TNF alpha level with concurrent reduced resistance to erythropoiesis stimulating agents (ESA) has been also reported with MCO-HD.

VieX (Polysulfone, surface area: 2.1 m², sterilization gamma, ultrafiltration coefficient: 104.3 ml/h/mmHg, Asahi Kasei Medical, Japan), a novel SHF vitamin E-coated dialyzer, which has larger pore size than HF dialyzer, might provide also higher middle molecules removal and more biocompatibility improvement.

Preliminary data demonstrate similar reduction ration of beta2-microglobulin, which is the most studied middle molecule, between MCO-HD and Super High Flux Vitamin E (SHFVE)-HD.

The aim of the present study was to compare the efficiency of the SHFVE dialyzer versus the MCO dialyzer on the removal of beta2-microglobulin and other middle molecules in a non-inferiority fashion, and their respective effects on inflammation, oxidative stress and biocompatibility parameters.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Age ≥ 18 years
* Patients established on HF-HD trice weekly four hour-sessions for at least 3 months

Exclusion Criteria:

* Malabsorption syndrome, active malignant disease or other critical illnesses and any ongoing condition that may interfere with inflammatory parameters (baseline C-Reactive Protein >40 mg/l)
* Pregnant or breast feeding women
* Any uncontrolled medical condition, psychiatric disorder or biological abnormality that might interfere with subject's participation or ability to sign an informed consent.
* Significant residual kidney function as defined by an urine output > 500 mL.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2023-06-14 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Beta2-microglobulin reduction ratio (RR) after 3 months of SHFVE-HD and MCO-HD in a non-inferiority fashion. | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Poitiers, Poitiers, France

REFERENCES:
- [Derived] Belmouaz M, Cogne E, Joly F, Duthe F, Desport E, Martin C, Hauet T, Giraud S, Lemarie E, Durocher L, Bridoux F. Effects of super high-flux vitamin E-coated and medium cut-off dialyzers on uremic toxins removal and biocompatibility: the E-FLUX randomized controlled study. Clin Kidney J. 2025 Apr 11;18(5):sfaf106. doi: 10.1093/ckj/sfaf106. eCollection 2025 May. PMID 40342620